CLINICAL TRIAL: NCT02331420
Title: Prospective Randomized Controlled Trial on the Effect of BAriatric Surgery Versus Optimal Medical Therapy on Cardiovascular Health and Progression of Atherosclerosis in Obese, Type II Diabetic Patients
Brief Title: Effect of BAriatric Surgery Versus Optimal Medical Therapy on Cardiovascular Health and Atherosclerosis in Obese, Type II Diabetic Patients
Acronym: BASTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Associate Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 4569/14
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Atherosclerosis
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Atherosclerosis | interventions — Gastric Bypass; Nutrition Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Bariatric Surgery (Experimental): Gastric bypass
  Interventions: Procedure: Gastric bypass
- Optimal Medical Therapy (Active Comparator): planned visits, optimized hypoglycemic treatment, diet and lifestyle modification
  Interventions: Behavioral: Medical therapy

INTERVENTIONS:
Procedure: Gastric bypass — A subcardial gastric pouch with a 30±10 ml capacity will be created by sectioning the stomach with a linear stapler 3-4 cm horizontally on the lesser curve, 4 cm distal to the e-g junction, and then vertically until attainment of the angle of Hiss. After identification of the Treitz ligament, the jejunum will be transected at 100 cm from the ligament of Treitz and the two stumps will be closed. The distal stump will be anastomosed to the distal end of the gastric pouch. The preferred gastro-jejunal anastomosis is the totally hand-sewn one, but it can be performed using any other the technique the surgeon is more familiar with. Finally, the proximal stump of the transacted bowel will be joined end-to-side to the jejunum 150 cm distal to the gastro-enterostomy.
  Arms: Bariatric Surgery
Behavioral: Medical therapy — * Assessment and treatment by a multidisciplinary team (diabetologist, dietitian, nurse);
  * Planned visits at baseline and at 1, 3, 6, 9, 12, and 24 months after study entry;
  * Oral hypoglycemic agents and insulin doses optimized on an individual basis with the aim of reaching a glycated hemoglobin level of less than 7%;
  * Programs for diet and lifestyle modification, including reduced overall energy and fat intake (<30% total fat, <10% saturated fat, and high fiber content) and increased physical exercise (≥30 minutes of brisk walking every day, possibly associated with moderate-intensity aerobic activity twice a week);
  * low-calorie diet (every day: 50% carbohydrate, 30% protein and 20% lipids).
  Arms: Optimal Medical Therapy

SUMMARY:
To assess the impact of weight loss due to bariatric surgery, as compared to the effect of optimal medical therapy alone on endothelial function, subclinical atherosclerosis, cardiovascular autonomic function in obese patient affected by type 2 diabetes.The study consists in a 2-arm randomized trial, in which patients will be randomly assigned to bariatric surgery or optimal medical therapy. Each patient will be studied at baseline (T0) and 12 months thereafter (T1).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes: the American Diabetes Association (ADA) recommends the following criteria for diagnosis of diabetes: HbA1c ≥6.5% OR fasting plasma glucose‡ ≥126 mg/dL (7.0 mmol/L) OR 2-hour plasma glucose ≥200 mg/dL (11.1 mmol/L) during an oral glucose tolerance test; 75-g glucose load should be used OR random plasma glucose concentration ≥200 mg/dL (11.1 mmol/L) in persons with symptoms of hyperglycemia or hyperglycemic crisis;
* indication to bariatric surgery: BMI ≥35 kg/m2 and one or more obesity related co-morbidities, including Type 2 Diabetes Mellitus.

Exclusion Criteria:

* overt cardiovascular disease (as assessed by clinical evaluation, physical examination, 12-lead ECG, 2D-echocardiogram);
* smoking habit;
* associated medical conditions, as chronic kidney disease (defined as creatinine clearance <60 mL/min/L.73m2), liver cirrhosis, malignancies, chronic congestive heart failure, acute or chronic inflammatory disease;
* specific contraindication to bariatric surgery;
* pregnancy;
* medical conditions requiring acute hospitalization;
* psychological conditions which may hamper patient's cooperation;
* geographic inaccessibility.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Subclinical Atherosclerosis (ecographic assessment of carotid artery intima-media thickness) | 12 months
  ecographic assessment of carotid artery intima-media thickness
Endothelial Function (ecographic assessment of flow-mediated dilation and nitrate mediated dilation) | 12 months
  ecographic assessment of flow-mediated dilation and nitrate mediated dilation
Cardiac autonomic function (heart rate variability measurements on 24-hour Holter ECG recordings) | 12 months
  heart rate variability measurements on 24-hour Holter ECG recordings